CLINICAL TRIAL: NCT03958760
Title: Characteristics, Treatment, and Economic Burden of Disease of Chinese Diabetic/Non-diabetic Patients With/Without Established Cardiovascular Disease, Chronic Kidney Disease, or at High Cardiovascular Risk
Brief Title: Characteristics, Treatment, and Economic Burden of Patients With CVD,CKD or at High Cardiovascular Risk
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Sun Xin, Professor, West China Hospital
Other Study IDs: CREAT-DIABETES
Record Dates: First submitted 2019-04-22; First posted 2019-05-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Cardiovascular Abnormalities; Chronic Kidney Diseases; Diabetes
MeSH Terms: conditions — Cardiovascular Abnormalities; Renal Insufficiency, Chronic; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Diabetic patients with CVD, CKD or at risk: The group A include all diabetic patients with established cardiovascular disease, chronic kidney disease, or at high cardiovascular risk.
- Diabetic patients without CVD, CKD or at risk: The group B include all diabetic patients without established cardiovascular disease, chronic kidney disease, or at high cardiovascular risk.
- Non-diabetic patients with CVD, CKD or at risk: The group C included all non-diabetic patients with established cardiovascular disease, chronic kidney disease, or at high cardiovascular risk.
- Health controls: The group D included non-diabetic patients without established cardiovascular disease, chronic kidney disease, and not at high cardiovascular risk.

SUMMARY:
The heavy disease burden is mainly due to diabetic complications. Diabetes is a major risk factor for cardiovascular disease (CVD) and chronic kidney disease (CKD).China has been the largest absolute disease burden of diabetes in the world recently1. Diabetic patients with established CVD or CKD are bringing growing pressure upon our nation's healthcare expenditure1. However, the characteristic profile of Chinese diabetic patients who has CVD, CKD or at high risk of CVD remains unclear thus is in urgent need for in-depth investigation.In current China, however, the information regarding diabetes or non-diabetes patients who also had other comorbid conditions (e.g. established CV diseases, CKD or at high risk for such problem), is limited; the patient characteristics, treatment patterns and economic burden may not be fully understood.Therefore, based on TianJin regional database, the investigators will describe the demographic, clinical characteristics, treatment, and economic burden of disease of Chinese diabetic/non-diabetic patients with/without established CV disease, CKD, or at high CV risk including hypertension and hyperlipidaemia. And the investigators believe that the resulting findings will inform a comprehensive group of evidence users to achieve better healthcare for diabetes patients with established or at high risk of CVD or CKD.

DETAILED DESCRIPTION:
The study aimed to investigate the clinical characteristics, treatment, and economic burden of disease of Chinese diabetic/non-diabetic patients with/without established cardiovascular disease, chronic kidney disease, or at high cardiovascular risk, including:

1. estimate the proportion of Chinese diabetic/non-diabetic patients with established cardiovascular disease, CKD, or at high cardiovascular risk including hypertension and hyperlipidaemia;
2. describe the demographic and clinical characteristics of Chinese diabetic/non-diabetic patients with/without established cardiovascular disease, CKD, or at high cardiovascular risk;
3. investigate the treatment patterns of Chinese diabetic/non-diabetic patients with/without established cardiovascular disease, CKD, or at high cardiovascular risk;
4. examine economic burden of disease of Chinese diabetic/non-diabetic patients with/without established cardiovascular disease, CKD, or at high cardiovascular risk;
5. explore the trends of clinical characteristics, treatment pattern, economic burden of inpatients over time (2008, 2013, and 2018 separately);

ELIGIBILITY:
Inclusion Criteria:

* Patients in the TianJin regional database from 2015 to 2018.
* patients with at least 1 discharged diagnosis or 2 outpatient diagnosis of ischemic heart diseases (ICD-10 I20~I25);
* patients with at least 1 discharged diagnosis or 2 outpatient diagnosis of cerebrovascular diseases (ICD-10 I60~I69);
* patients with at least 1 discharged diagnosis or 2 outpatient diagnosis of ischemic peripheral artery disease (ICD-10 E10.501, E11.603, E14.501, E14.606, E14.503, I73.9, I99.03, I99.04);
* patients with at least 1 discharged diagnosis or 2 outpatient diagnosis of heart failure (ICD-10 I50);
* inpatients with at least once 1 discharged diagnosis CKD (ICD-10 N18), or inpatients with the last estimated glomerular filtration rate (eGFR, calculated by CKD-EPI equation) <60 mL/min/1.73 m2 or prescription of dialysis, but not with the diagnosis of acute kidney injury (ICD-10 N17)
* Outpatients with at least 2 diagnosis of CKD or with two consecutive eGFR(calculated by CKD-EPI equation) <60 mL/min/1.73 m2 by 90 days or more.
* patients with at least 1 discharged diagnosis or 2 outpatient diagnosis of hypertension (ICD-10 I10~I15);
* at least 1 discharged diagnosis or 2 outpatient diagnosis of hyperlipidaemia (ICD-10 E78.001-E78.003, E78.101, E78.203, E78.301-E78.304, E78.306, E78.401, E78.501, E78.902)
* patients with at least 1 discharged diagnosis or 2 outpatient diagnosis of diabetes (ICD-10 E10-E14)
* In addition, we will randomly select a group of non-diabetic patients without any of the above diseases by matching on age and gender.

Exclusion Criteria:

* Patients with non-Chinese nationalities;
* Patients with abnormal bill (planning to define abnormal bill as the top 1-2.5% of total medical costs in three groups, respectively, but the final standard will be defined based on the real extracted data);
* Duplicated storage (records with same inpatient code).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetic/non-diabetic patients with/without established cardiovascular disease, chronic kidney disease, or at high cardiovascular risk in TianJin regional database
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
The number of diabetic/non-diabetic patients with disease or risk | 10 months after enrollment
  The number of diabetic patients with established cardiovascular disease, chronic kidney disease, or at high cardiovascular risk among all patients with diabetes;
The proportion of diabetic/non-diabetic patients with disease or risk | 10 months after enrollment
  The proportion of diabetic/non-diabetic patients with established cardiovascular disease, chronic kidney disease, or at high cardiovascular risk among patients without diabetes
The demographic characteristics of the last visit for all patients of the studied population | 10 months after enrollment
  1. age at admission;
  2. gender;
  3. ethnic;
  4. insurance payment;
The diagnosis of patients | 10 months after enrollment
  The number of patients with diagnosis at the last visit
The proportion of death | 10 months after enrollment
  The proportion of death at the last visit; the proportion of death at admission of the last visit for inpatients in 2008, 2013 and 2018.
Random blood glucose (mmol/L) | 12 months after enrollment
  The most recent value of random blood glucose (mmol/L) within the previous year for outpatients; the value of random blood glucose (mmol/L) at admission of the last visit for inpatients in 2008, 2013, 2018.
HbA1C (%) | 12 months after enrollment
  The most recent value of HbA1C (%) within the previous year for outpatients; the value of HbA1C (%) at admission of the last visit for inpatients in 2008, 2013, 2018.
Department of discharge for hospitalized patients | 12 months after enrollment
  Department of discharge of the last visit for hospitalized patients; and summarize the number of patients of different department of discharge in 2008, 2013, 2018.
serum creatinine (μmol/L) | 12 months after enrollment
  The most recent value of serum creatinine (μmol/L) within the previous year for outpatients; the value of serum creatinine (μmol/L) at admission of the last visit for inpatients in 2008, 2013, 2018.
eGFR (mL/min/1.73m2) | 12 months after enrollment
  The most recent value of eGFR (mL/min/1.73m2) within the previous year for outpatients; the value of eGFR (mL/min/1.73m2) at admission of the last visit for inpatients in 2008, 2013, 2018.
Microalbuminuria (MALB) (mg/24h) | 12 months after enrollment
  The most recent value of microalbuminuria (MALB, mg/24h) within the previous year for outpatients; the value of microalbuminuria (MALB, mg/24h) at admission of the last visit for inpatients in 2008, 2013, 2018.
High density lipoprotein (HDL) (mmol/L) | 12 months after enrollment
  The lasted examination of high density lipoprotein (HDL) (mmol/L) within the last year for outpatients; the value of high density lipoprotein (HDL) (mmol/L) at admission of the last visit for inpatients in 2008, 2013, 2018.
Low density lipoprotein (LDL) (mmol/L) | 12 months after enrollment
  The lasted examination of low density lipoprotein (HDL) (mmol/L) within the last year for outpatients; the value of low density lipoprotein (HDL) (mmol/L) at admission of the last visit for inpatients in 2008, 2013, 2018.
Total cholesterol (TC) (mmol/L) | 12 months after enrollment
  The lasted examination of total cholesterol (TC) (mmol/L) within the last year for outpatients; the value of total cholesterol (TC) (mmol/L) at admission of the last visit for inpatients in 2008, 2013, 2018.
Triglyceride (TG) (mmol/L) | 12 months after enrollment
  The lasted examination of triglyceride (TG) (mmol/L) within the last year for outpatients; the value of triglyceride (TG) (mmol/L) at admission of the last visit for inpatients in 2008, 2013, 2018.

SECONDARY OUTCOMES:
The number of patients with different treatment pattern | 10 months after enrollment
  1. number of patients with the treatment of antiplatelet drug,statin,vasodilators.
  2. number of patients with the treatment of different insulin and OHA prescription;
  3. number of patients with the treatment of anti-hypertensive drugs (CCB, ACEI/ARB, beta-blocker and diuretic)
  4. number of patients with the treatment of statin and fibrates;
  5. number of patients with the treatment of the dialysis, ACEI/ARB and the kindney transplantation.
  We descirbe the treatment pattern based on treatment prescribed during the most recent visit for all inpatients, and based on at least 2 prescription within the previous year for outpatients
The length of stay in the hospital | 12 months after enrollment
  describe the length of stay in the hospital of the last hospitalization, the length stay in the hospital for inpatients from 2008 to 2018.
The economic burden | 12 months after enrollment
  hospitalization cost of the studied population for the last visit; total cost and hospitalization cost of the studied population from 2008 to 2018.
Numbers of admissions | 12 months after enrollment
  The total number of admissions for inpatients from 2008 to 2018
The proportion of re-hospitalization | 12 months after enrollment
  The last visiting and previous one within 30 days and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, PhD, Study Director — The West China Hospital of Sichuan university
Locations (1):
- Tian Jin Healthcare Big Data Co. Ltd, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No